CLINICAL TRIAL: NCT06874374
Title: Closed-Loop Transcranial Alternating Current Stimulation (CL-tACS) for the Treatment of Major Depressive Disorder: Double-Blind, Sham-Controlled Randomized Pilot Study
Brief Title: Individualized Non-invasive Brain Stimulation for the Treatment of Major Depressive Disorder
Acronym: CL-tACS RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulvinar Neuro, LLC (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: 24-2166; R44MH119872 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-03-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Depression - Major Depressive Disorder; Transcranial Alternating Current Stimulation
Keywords: tACS; Depression; Major Depressive Disorder; Transcranial Alternating Current Stimulation
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Closed-loop tACS (Experimental): Closed-loop individual alpha tACS daily for five consecutive days.
  Interventions: Device: Closed-loop tACS
- Sham Closed-loop tACS (Sham Comparator): Sham closed-loop individual alpha tACS daily for five consecutive days.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Closed-loop tACS — Individual alpha tACS
  Other Names: CL-tACS
  Arms: Active Closed-loop tACS
Device: Sham Comparator — Sham stimulation
  Arms: Sham Closed-loop tACS

SUMMARY:
The purpose of this research study is to study a closed-loop transcranial alternating current stimulation (tACS) device to evaluate feasibility of the product in a clinical trial and collect preliminary data on potential effects on symptoms of depression in people with major depressive disorder.

DETAILED DESCRIPTION:
The purpose of this study is to investigate device feasibility and performance of the XCSITE 100 Pro V2 device and assess preliminary efficacy of closed-loop transcranial alternating current stimulation (CL-tACS) for reducing symptoms of major depressive disorder (MDD) in a double-blind, sham-controlled, parallel group, single-site clinical trial. A total of 40 participants will be randomized to receive active or sham CL-tACS via carbon-silicone electrodes for up to 40 minutes over 5 consecutive days. Device feasibility and performance data will be collected from every stimulation session. Clinical assessments of depression and related symptoms will be performed at Baseline (Day 1), End Of Treatment (EOT; Day 5), and Follow-Up (FUP, 2-weeks post-treatment, Day 19). High-density electroencephalography (HD-EEG) will be performed at Baseline, EOT and FUP. An optional MRI will be performed up to 30 days before, or on Baseline, to provide anatomical data for EEG brain connectivity analysis.

ELIGIBILITY:
Inclusion Criteria:

* Any gender, aged 18 - 70
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* DSM-5 diagnosis of unipolar, non-psychotic MDD as evidenced by the DIAMOND
* HDRS-17 score ≥14
* Low suicide risk (defined for this study as no active suicidal ideation in the past month and no suicide attempts, preparatory actions, or significant non-suicidal self-harm in the previous 2 years). Risk will be assessed utilizing the C-SSRS screen and triage version with further exploration of positive responses.
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* For people of childbearing potential: use of highly effective contraception as determined by the Investigator for at least 1 month prior to screening and agreement to use such a method during study participation

Exclusion Criteria:

* DSM-5 diagnosis of severe alcohol use disorder (AUD) within the last 12 months, as evidenced by the DIAMOND
* DSM-5 diagnosis of moderate to severe substance use disorder (excluding tobacco) within the last 12 months, as evidenced by the DIAMOND
* Lifetime history of bipolar disorder, as evidenced by DIAMOND
* Schizophrenia spectrum and other psychotic disorders, as evidenced by DIAMOND
* History of autism spectrum disorder
* Initiated any new psychotropic medication in the 6 weeks prior to screening or had a dose change in the preceding 6 weeks
* Initiated a new course of psychotherapy in the 6 weeks preceding screening
* Received any neurostimulation treatment in the 6 weeks preceding screening
* History of seizures (excluding febrile seizures in childhood or Electroconvulsive Therapy (ECT) induced seizures)
* Neurological disorders that would increase risk of participation or present a significant confounder in the opinion of the investigator (for example, dementia, history of stroke, Parkinson's disease, multiple sclerosis, history of traumatic brain injury with prolonged loss of consciousness, ruptured cerebral aneurysm, previous CNS radiation)
* Previously failed to respond to ECT or transcranial magnetic stimulation (TMS)
* Prior brain surgery and/or brain implants
* Implanted medical device that uses electricity
* Current pregnancy or lactation
* Currently enrolled in another clinical trial for depression
* For the optional MRI session only: Contraindication to MRI according to MRI Screening Form
* Unstable medical disorder or anything that would place the participant at increased risk or preclude the participant's full compliance with or completion of the study, in the opinion of the Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Correct Assignment by Device of Study Arm | 5 days
  Successful assignment by device software to correct study arm for each participant for each session, Day 1 (D1) through Day 5 (D5). Measured as percentage of successful assignments compared to intended programming.
Accuracy of Device Study Arm Parameters by Device | 5 days
  Verification of correct study arm parameters applied by device for each participant for each session, Day 1 (D1) through Day 5 (D5).
Accuracy of Stimulation Initiation Based on EEG by Device | 5 days
  Verification of correct stimulation initiation decisions for each evaluated EEG window by device for each participant for each session, Day 1 (D1) through Day 5 (D5).
Accuracy of Device Logs Uploaded to Cloud by Device | 5 days
  Verification of equivalence between logs stored on local device and corresponding logs uploaded to cloud for each participant for each session, Day 1 (D1) through Day 5 (D5).

SECONDARY OUTCOMES:
HDRS-17 Change | 21 Days
  Change in HDRS-17 from two week follow-up (FUP) to D1 between Experimental and Sham Comparator study arms; minimum value is 0, maximum value is 52. Higher scores indicate worse outcome.
Change in Alpha Oscillation Power | 5 Days
  Change in EEG alpha oscillation power between D1 and D5 between Experimental and Sham Comparator study arms.

OTHER OUTCOMES:
Change in Alpha Oscillation Power and Connectivity | 21 Days
  Change in HD-EEG alpha oscillation power and connectivity at D1, D5, and FUP between Experimental and Sham Comparator study arms.
Remission Rate | 21 Days
  Difference in remission rates between Experimental and Sham Comparator study arms at FUP. Remission defined as HDRS-17 score of less than or equal to 7.
Response Rate | 21 Days
  Difference in response rates between Experimental and Sham Comparator study arms at FUP. Response defined as greater than or equal to 50% reduction in HDRS-17 score from D1 to FUP.
SSRI Effect on HDRS-17 Change | 21 Days
  Change in HDRS-17 for Experimental study arm from two week follow-up (FUP) to D1 between patients on SSRI medication and patients not on SSRI medication; minimum value is 0, maximum value is 52. Higher scores indicate worse outcome.
Change in Quick Inventory of Depressive Symptomatology (QIDS) | 21 Days
  Change in QIDS from D1 to FUP between Experimental and Sham Comparator study arms; minimum value is 0, maximum value is 27. Higher scores indicate worse outcome.
Change in Snaith-Hamilton Pleasure Scale (SHAPS) | 21 Days
  Change in SHAPS from D1 to FUP between Experimental and Sham Comparator study arms; minimum value is 0, maximum value is 14. Higher scores indicate worse outcome.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire, short form (Q-LES-Q-SF) | 21 Days
  Change in Q-LES-Q-SF from D1 to FUP between Experimental and Sham Comparator study arms; minimum value is 0, maximum value is 14. Higher scores indicate worse outcome.
Change in Clinical Global Impression Scale (CGI) | 21 Days
  Change in CGI from D1 to FUP between Experimental and Sham Comparator study arms; CGI scale contains two scoring components, 1) Severity of Illness (0-7) and 2) Global Improvement (0-7). Higher scores in component 1 indicate worse symptoms while higher numbers in component 2 indicate worse clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: David Rubinow, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schwippel T, Pupillo F, Feldman Z, Walker C, Townsend L, Rubinow D, Frohlich F. Closed-Loop Transcranial Alternating Current Stimulation for the Treatment of Major Depressive Disorder: An Open-Label Pilot Study. Am J Psychiatry. 2024 Sep 1;181(9):842-845. doi: 10.1176/appi.ajp.20230838. Epub 2024 Aug 7. No abstract available. PMID 39108159
- [Background] Alexander ML, Alagapan S, Lugo CE, Mellin JM, Lustenberger C, Rubinow DR, Frohlich F. Double-blind, randomized pilot clinical trial targeting alpha oscillations with transcranial alternating current stimulation (tACS) for the treatment of major depressive disorder (MDD). Transl Psychiatry. 2019 Mar 5;9(1):106. doi: 10.1038/s41398-019-0439-0. PMID 30837453